CLINICAL TRIAL: NCT07154732
Title: Transcranial Photobiomodulation With Multiple Interventions in Children With Attention-Deficit/Hyperactivity Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QL000006
Record Dates: First submitted 2025-07-20; First posted 2025-09-04 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: transcranial Light Stimulation (tLS); transcranial photobiomodulation (tPBM); Attention Deficit Hyperactivity Disorder (ADHD); Electroencephalography (EEG)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tPBM session (Active Comparator): During the active stimulation period, participants completed 11 sessions of active stimulation within 11 days in their own homes. The stimulation duration per session was 9-12 minutes, administered once daily.
  Interventions: Device: Transcranial photobiomodulation (active)
- Sham tPBM session (Sham Comparator): During the sham stimulation period, participants completed 11 sessions of sham stimulation in their own homes within 11 days, with the same stimulation frequency and duration as the active stimulation group. The intervention was delivered at the same target area and wavelength; the intensity was matched to that of the active stimulation during the first 30 seconds and the last 30 seconds of each session, while no intervention was applied in the intermediate period.
  Interventions: Device: Transcranial photobiomodulation (sham)

INTERVENTIONS:
Device: Transcranial photobiomodulation (active) — During the active stimulation period, participants completed 11 sessions of active stimulation within 11 days in their own homes. The stimulation duration per session was 9-12 minutes, administered once daily.
  Arms: Active tPBM session
Device: Transcranial photobiomodulation (sham) — During the sham stimulation period, participants completed 11 sessions of sham stimulation in their own homes within 11 days, with the same stimulation frequency and duration as the active stimulation group. The intervention was delivered at the same target area and wavelength; the intensity was matched to that of the active stimulation during the first 30 seconds and the last 30 seconds of each session, while no intervention was applied in the intermediate period.
  Arms: Sham tPBM session

SUMMARY:
To investigate the therapeutic efficacy of transcranial photobiomodulation (tPBM) with multiple interventions in children and adolescents with attention-deficit/hyperactivity disorder (ADHD). The study evaluates intervention effects at Magnetic Resonance Imaging, electrophysiological, Visual Search Task, cognitive-behavioral, and clinical symptom levels, aiming to identify the optimal clinical treatment regimen for ADHD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6 and 18 years;
2. Clinically diagnosed with ADHD by a psychiatrist;
3. Confirmed by the researcher (child psychiatrist) to meet the diagnostic criteria for Attention-Deficit/Hyperactivity Disorder as outlined in the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5);
4. M.I.N.I. KID interview shows only ADHD, with no other comorbidities;
5. Able to cooperate with transcranial photobiomodulation.
6. The participant and their guardian fully understand the study procedures and content and agree to participate in the study, signing the informed consent form.

Exclusion Criteria:

1. Diagnosis of other severe mental illnesses, such as schizophrenia or bipolar disorder;
2. Presence of severe physical diseases or conditions, such as significant intracranial lesions, thyroid disorders, epilepsy, congenital heart disease, severe hematologic disorders, systemic lupus erythematosus, auditory or visual impairments, etc.;
3. Presence of significant structural brain abnormalities on imaging studies;
4. Presence of severe neurological diseases with a clear family history or potential risk;
5. Presence of metal implants or a pacemaker, or holes or fractures in the skull;
6. Currently undergoing other ADHD treatments (e.g., methylphenidate or other pharmacological treatments, behavioral therapy, etc.) or has discontinued such treatments for less than 2 weeks;
7. Raven's Progressive Matrices IQ score < 85.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Swanson, Nolan, and Pelham Version IV(SNAP-IV) | From enrollment to one week after the end of the second group's intervention.
  The Swanson, Nolan, and Pelham Version IV (SNAP-IV) scale includes a total score and three subset scores, with higher scores indicating more severe ADHD symptoms.
Sleep Disturbances Scale for Children(SDSC) | From enrollment to one week after the end of the second group's intervention.
  The Sleep Disturbances Scale for Children (SDSC) is a widely used standardized tool designed to assess sleep problems in children and adolescents (typically aged 6-18 years). It evaluates various dimensions of sleep disturbances, with subscales (subsets) that target specific types of sleep disorders. Higher scores indicate more prominent sleep problems.
Behavioral Inhibition/Activation System Scales (BIS/BAS) | From enrollment to one week after the end of the second group's intervention.
  The Behavioral Inhibition/Activation System Scales (BIS/BAS) is a widely used self-report instrument designed to assess individual differences in two fundamental motivational systems proposed by Gray's reinforcement sensitivity theory: the Behavioral Inhibition System (BIS) and the Behavioral Activation System (BAS). High BIS scores: Indicate a heightened sensitivity to negative stimuli, punishment, or potential threats. BAS scores primarily reflect sensitivity to positive stimuli/rewards: Higher scores = greater motivation, impulsivity, or approach behavior; lower scores = reduced reward responsiveness or motivation. The BAS scale typically includes three subscales.

SECONDARY OUTCOMES:
EEG(Electroencephalogram) | From enrollment to one week after the end of the second group's intervention.
  Electroencephalogram (EEG) was recorded during participants' performance of a visual search task. The primary analyses focused on the latency and amplitude of the N2pc waveform, as well as the power spectra of bands such as alpha, during the task performance both before and after the intervention.
Executive Function Task | From enrollment to one week after the end of the second group's intervention.
  Participants completed an executive function task following active and sham stimuli to compare the effects of transcranial light stimulation(tLS) on the improvement of executive function in children with ADHD.
Visual Search Task | From enrollment to one week after the end of the second group's intervention.
  At the start of the task, participants were required to fixate on the central fixation point on the screen. Subsequently, a search matrix was presented briefly before disappearing. Participants needed to judge the location of the target, move the joystick, and press the confirmation button to terminate the trial.
Photobiomodulation Subjective Assessment Scale | From enrollment to one week after the end of the second group's intervention.
Magnetic Resonance Imaging | From enrollment to one week after the end of the second group's intervention.
  Participants underwent magnetic resonance imaging scans before and after the interventions in both groups to clarify the intervention effects of the active and sham stimulus groups.